CLINICAL TRIAL: NCT02301416
Title: Qsymia as an Adjunct to Surgical Therapy in the Superobese
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00027047
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-11

CONDITIONS: Obesity; Metabolic Surgery; Weight Loss; Bariatric Surgery Procedures
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Qsymia; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentermine/topiramate (Experimental): All subjects enrolled in the study will be placed on the study medication.
  Interventions: Drug: Phentermine/topiramate; Other: low calorie diet
- Historical Control (No Intervention): Historical controls who had sleeve gastrectomy during the same time frame without phentermine/topiramate treatment

INTERVENTIONS:
Drug: Phentermine/topiramate — Minimum of 3 months on Qsymia (7.5/46 mg) prior to scheduled weight loss surgery and continuance of up to 24 months of Qsymia after scheduled weight loss surgery.
  Other Names: Qsymia
  Arms: Phentermine/topiramate
Other: low calorie diet — The low-calorie diet will be individually tailored based on initial resting metabolic rate measurement and co-morbid conditions.
  Arms: Phentermine/topiramate

SUMMARY:
This study tests the efficacy of the medication, Qsymia, as an adjunct therapy in superobese individuals planning to undergo weight loss surgery. Individuals taking the medication before and after surgery will be compared to historical controls who had surgery without taking the medication.

DETAILED DESCRIPTION:
While there is obvious focus on the obesity epidemic that affects approximately one-third of the U.S. population, one subgroup within the epidemic remains on the fringe of scientific study and effective treatment options. The super obese patient, in this instance defined as those with a BMI ≥ 50 kg/m2, presents a difficult treatment challenge in managing this level of obesity. While bariatric surgery, including Roux-en-Y gastric bypass and biliopancreatic diversion with duodenal switch, have been shown to be effective in severe obesity (BMI ≥ 40 kg/m2), the risks involved with surgical intervention in the super obese patient are high.

Qsymia provides a potential opportunity to develop an effective treatment plan that would be an adjunct to surgical intervention in the super obese patient. Use of Qsymia in addition to a low-calorie dietary prescription pre-operatively would effectively decrease weight prior to surgical intervention, lowering surgical risk to some extent. Additionally, if continued post-operatively, Qsymia as an adjunct to the post-surgical dietary plan would potentially extend the weight loss horizon so that the probability of the typical weight loss plateau at 12-18 months is decreased.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 50 kg/m2
* Determined to be a good candidate for surgery based on medical and psychological exam.
* Willing to participate in a 3-6 month medically supervised weight loss plan prior to surgery.
* Planning to remain in the reasonable vicinity of the Wake Forest Baptist Health - Weight Management Center for the duration of the study.

Exclusion Criteria:

* History of prior weight loss surgery (removal/conversion from band to sleeve will not be excluded)
* Pregnant (women of childbearing potential will complete a pregnancy test (blood draw) to make sure they are not pregnant at the time that they initiate the medication). Ongoing monitoring of pregnancy status is the responsibility of the patient and they are instructed as such in the consent form.
* Ongoing use of weight loss medication
* Contraindications to use of Qsymia, including pregnancy, history of glaucoma, unstable cardiac disease (unstable angina, recent heart attack or stroke (in the past 6 months), uncontrolled arrhythmia), hyperthyroidism, taking monoamine oxidase inhibitors (MAOIs) or allergy to either topiramate or sympathomimetic amines like phentermine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamy D Ard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective chart review patients were not considered enrolled, but historical data was used as a comparison so it is included.
Groups:
- Historical Control: Retrospective chart review of patients who had sleeve gastrectomy without phentermine/topiramate
Period: Overall Study
Arm/Group | Phentermine/Topiramate | Historical Control
Started | 25 | 40
Completed | 15 | 40
Not Completed | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surgery Only: Historical controls who had sleeve gastrectomy without phentermine/topiramate
- Total: Total of all reporting groups
Arm/Group | Phentermine/Topiramate | Surgery Only | Total
Number analyzed (Participants) | 15 | 40 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (7.3) | 45 (10.8) | 44.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 33 | 45
  Male | 3 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 40 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 03 | 9 | 12
  White | 12 | 31 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 40 | 55
Body weight [Mean (Standard Deviation); unit: kilograms] | 178.9 (31.1) | 159.5 (21) | 164.8 (25.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 61.2 (7.1) | 57 (5.6) | 58.1 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who do Not Meet the Criteria to Move Forward With Roux en Y Gastric Bypass (RYGB)
Description: Proportion of patients who do not meet the criteria to move forward with a second surgical procedure following an initial procedure plus the medication Qsymia. The criteria that suggest RYGB is indicated are: 1) BMI of 40 or greater or 2) BMI of 35-39.9 with poorly controlled co-morbidities.
Time Frame: 24 months post-operatively
Population: 2 participants had RYGB instead of Sleeve Gastrectomy
Measure: Count of Participants; unit: Participants
Groups:
- Surgery Only: Historical controls who had surgery only
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
Participants | 8 | 19

2. Secondary Outcome: Percent Weight Change
Description: Percent weight loss achieved before and after surgery while taking the medication, Qsymia.
Time Frame: Pre-operatively and 24 months post-operatively
Population: 2 participants had RYGB instead of sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: Percentage of weight change
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
Percentage of weight change | -38.16 [-45.39 to -30.94] | -27 [-31.02 to -22.99]

3. Secondary Outcome: Body Mass Index
Description: Resulting body mass index
Time Frame: 24 months post-operatively
Population: 2 participants had RYGB instead of Sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
kg/m^2 | 33.79 [29.47 to 38.12] | 41.96 [39.47 to 44.45]

4. Secondary Outcome: Percent Body Fat
Description: Change in percent body fat
Time Frame: 24 months post-operatively
Population: Measure not obtained
Arm/Group | Phentermine/Topiramate | Historical Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate via indirect calorimetry
Time Frame: 24 months post-operatively
Population: Outcome measure not obtained
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percent Weight Change
Description: Percent weight loss achieved before and after surgery while taking the medication, Qsymia.
Time Frame: Pre-operatively and 12 months post-operatively
Population: 2 participants had RYGB instead of sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
Percent | -39.34 [-45.36 to -33.32] | -31.43 [-34.86 to -28.01]

7. Secondary Outcome: Percent Weight Change
Description: Percent weight loss achieved before and after surgery while taking the medication, Qsymia.
Time Frame: Pre-operatively and 6 months post-operatively
Population: 2 participants had RYGB instead of sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
Percent | -32.79 [-37.56 to -28.02] | -27.25 [-29.97 to -24.53]

8. Secondary Outcome: Percent Weight Change
Description: Percent weight loss achieved before and after surgery while taking the medication, Qsymia.
Time Frame: Pre-operatively and 3 months post-operatively
Population: 2 participants had RYGB instead of sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
Percent | -25.24 [-29.63 to -20.84] | -21.46 [-23.96 to -18.97]

9. Secondary Outcome: Body Mass Index
Description: Resulting body mass index
Time Frame: 12 months post-operatively
Population: 2 participants had RYGB instead of Sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
kg/m^2 | 33.46 [29.94 to 36.98] | 39.53 [37.43 to 41.63]

10. Secondary Outcome: Body Mass Index
Description: Resulting body mass index
Time Frame: 6 months post-operatively
Population: 2 participants had RYGB instead of Sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
kg/m^2 | 37.61 [34.83 to 40.38] | 41.93 [40.23 to 43.63]

11. Secondary Outcome: Body Mass Index
Description: Resulting body mass index
Time Frame: 3 months post-operatively
Population: 2 participants had RYGB instead of Sleeve gastrectomy
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 13 | 40
kg/m^2 | 42.31 [39.78 to 44.84] | 45.28 [43.71 to 46.84]

12. Secondary Outcome: Percent Body Fat
Description: Change in percent body fat
Time Frame: 12 months post-operatively
Population: Measure not obtained
Arm/Group | Phentermine/Topiramate | Historical Control
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percent Body Fat
Description: Change in percent body fat
Time Frame: 6 months post-operatively
Population: Measure not obtained
Arm/Group | Phentermine/Topiramate | Historical Control
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percent Body Fat
Description: Change in percent body fat
Time Frame: 3 months post-operatively
Population: Measure not obtained
Arm/Group | Phentermine/Topiramate | Historical Control
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate via indirect calorimetry
Time Frame: 12 months post-operatively
Population: Outcome measure not obtained
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate via indirect calorimetry
Time Frame: 6 months post-operatively
Population: Outcome measure not obtained
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate via indirect calorimetry
Time Frame: 3 months post-operatively
Population: Outcome measure not obtained
Arm/Group | Phentermine/Topiramate | Surgery Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events ascertained at each clinical follow up. Retrospective chart review patients were not considered enrolled, so adverse event information was not collected for them.
Arm/Group | Phentermine/Topiramate
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 3/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phentermine/Topiramate (N=25)
Panniculitis (Infections and infestations) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phentermine/Topiramate (N=25)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
insomnia (Nervous system disorders) | 1 (1)
irritability (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an open-label, nonrandomized observational trial of only 2 years postoperative follow-up.

We also did not control for the amount of contact that patients received in the course of their treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02301416/Prot_SAP_000.pdf